CLINICAL TRIAL: NCT01201668
Title: Persistent Pain and Root Canal Therapy
Brief Title: DPBRN Persistent Pain and Root Canal Therapy
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other); University of Copenhagen (Other); University of Florida (Other); University of Alabama at Birmingham (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Gregg H. Gilbert, DDS, MBA, FAAHD, Professor and Chair, Department of General Dental Sciences, Dental Practice-Based Research Network
Other Study IDs: 133265; U01DE016747 (NIH)
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Root Canal Therapy; Persistent Tooth Pain
Keywords: post-operative pain; root canal therapy; feasibility; post-surgical persistent pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Persistent Tooth Pain

SUMMARY:
The purpose of this study is to document by survey the occurence of tooth pain present 3 months and 6 months after root canal therapy in the patients recruited for the DPBRN "Peri-operative tooth pain" study. This study will access the feasibility of obtaining 3 month and 6 month follow-up data on the patient enrolled in the DPBRN "Peri-operative tooth pain" study.

ELIGIBILITY:
Inclusion Criteria:

* 19-70 years old
* Permanent adult tooth requiring its first non-surgical root canal therapy
* patients with more than 1 tooth requiring root canal therapy are eligible, but only the first root canal procedure will be included to avoid problems of correlation within patients

Exclusion Criteria:

* evidence of prior root canal therapy, including iatrogenic, but not disease-induced pulp access of the tooth being considered
* patients with obvious cognitive impairments (e.g., past stroke with communication deficits, dementia,mental disability)
* patients unable to return for 6 month follow-up

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants directly involved in this study are the patients who have sought dental treament in the practitioner-investigators' practices. The practitioner-investigators will be endodontists and general dentists.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Nixdorf, DDS, MS, Principal Investigator — University of Minnesota
Locations (8):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida College of Dentistry, Gainesville, Florida
  - Health Partners Dental Group, Minneapolis, Minnesota
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Permanente Denrtal Associates, Portland, Oregon
- University of Copenhagen Royal Dental College, Copenhagen, Denmark

REFERENCES:
- See also: Dental Practice-Based Research Network — http://DentalPBRN.org
- See also: Dental Practice-Based Research Network — http://DPBRN.org